CLINICAL TRIAL: NCT03086668
Title: Tube-Videostylet Assembly for Nasotracheal Intubation Assisted by a Fingers-Hook Technique
Brief Title: Fingers Hook Technique to Facilitate Nasotracheal Intubation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: KMUHIRB-E(I)-20160019
Record Dates: First submitted 2017-02-01; First posted 2017-03-22 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2018-08

CONDITIONS: Nasotracheal Intubation
Keywords: Nasotracheal Intubation; jaw thrust; hook-finger

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Jaw thrust Group (Experimental): an assembly of video-stylet and double curve endotracheal tube with conventional jaw thrust technique to facilitate nasotracheal intubation
  Interventions: Procedure: Conventional Jaw thrust Group
- Fingers hook Group (Experimental): an assembly of video-stylet and double curve endotracheal tube with fingers-hook technique to facilitate nasotracheal intubation
  Interventions: Procedure: Fingers hook Group

INTERVENTIONS:
Procedure: Conventional Jaw thrust Group — a video-stylet assisted nasotracheal intubation and facilitate by conventional jaw thrust technique
  Arms: Conventional Jaw thrust Group
Procedure: Fingers hook Group — a video-stylet assisted nasotracheal intubation and facilitate by fingers-hook technique
  Arms: Fingers hook Group

SUMMARY:
to compare either using conventional jaw thrust technique or with a novel fingers-hook technique to facilitate video-stylet assisted nasotracheal intubation

DETAILED DESCRIPTION:
It is necessary to adequately exposure of glottis during naso-tracheal intubation using video-stylet. However, inadequate upward epiglottis or over-elevation of arytenoids all inhibit the tube tip smoothly into trachea. Therefore, the study is to investigate either jaw thrust or fingers-hook technique is advantages of nasotracheal intubation.

ELIGIBILITY:
Criteria:

Inclusion Criteria:

1. patients with American Society of Anesthesiologists physical status I-III
2. aged 20-65 years
3. Requiring general anesthesia undergoing oxo-maxillofacial surgery
4. unlimited mouth open
5. unlimited neck motion

Exclusion Criteria:

1. mouth open < 3 cm
2. Ankylosing arthritis patients.
3. BMI≧35 kg/m2

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-03-27 (Actual); Primary Completion 2018-11-11 (Actual); Study Completion 2019-11-05 (Actual)

PRIMARY OUTCOMES:
grade of glottic field exposure and nasotracheal difficulty intubation score | half an hour
  to compare the two different techniques in glottic field exposure and score of nasotracheal difficulty intubations scale

SECONDARY OUTCOMES:
the tube-videostylet assembly range of motion | half an hour
  range motion of tip of tube-videostylet assembly advanced from nasal cavity to trachea

CONTACTS AND LOCATIONS:
Overall Officials: Kuang I Cheng, MD, PhD, Study Director — Department of Anesthesiology, Kaohsiung Medical University Hospital, Kaohsiung Medical University,Taiwan
Locations (1):
- Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung Medical University, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cheng KI, Yun MK, Chang MC, Lee KW, Huang SC, Tang CS, Chen CH. Fiberoptic bronchoscopic view change of laryngopharyngeal tissues by different airway supporting techniques: comparison of patients with and without open mouth limitation. J Clin Anesth. 2008 Dec;20(8):573-9. doi: 10.1016/j.jclinane.2008.01.013. PMID 19100929